CLINICAL TRIAL: NCT00909441
Title: Sentinel Node Biopsy Following NeoAdjuvant Chemotherapy in Biopsy Proven Node Positive Breast Cancer: A Multi-institutional Prospective Study Furthering the Treatment of Breast Cancer
Brief Title: Sentinel Node Biopsy Following NeoAdjuvant Chemotherapy in Biopsy Proven Node Positive Breast Cancer
Acronym: SN-FNAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Quebec Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE 08.224
Record Dates: First submitted 2009-05-25; First posted 2009-05-28 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2011-06

CONDITIONS: Breast Cancer; Invasive Breast Cancer
Keywords: Breast Cancer; Node Positive Breast Cancer; Sentinel Lymph Node Biopsy; Breast Surgery; Axillary Lymph Node Dissection; Neoadjuvant Chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SNB + ALND (Experimental): Intervention: Sentinel Lymph Node Biopsy followed by Axillary Node Dissection.
  Interventions: Procedure: Sentinel Lymph Node Biopsy

INTERVENTIONS:
Procedure: Sentinel Lymph Node Biopsy — Sentinel node biopsy is a technique in which a radioactive isotope is injected in the breast, with or without blue dye. These substances will then migrate and concentrate in the first nodes in the axilla that drain the breast: The sentinel nodes. These nodes (usually one to four nodes) are then evaluated for the presence of cancer cells.

SUMMARY:
Title of Study: Sentinel node biopsy following neoadjuvant chemotherapy in biopsy proven node positive breast cancer.

Objectives of the study:

Primary objective

1. Evaluate the accuracy of sentinel node biopsy in breast cancer patients presenting with positive nodal disease, proven by ultrasound guided fine needle aspiration, following neoadjuvant chemotherapy.

Secondary objectives

1. Evaluate the technical success of sentinel node biopsy following neoadjuvant chemotherapy.
2. Evaluate the accuracy of clinical examination and ultrasound examination of the axilla in identifying the presence of residual disease in the axilla following neoadjuvant chemotherapy in biopsy proven node positive breast cancer patients.

Number of patients:

N = 300

Population:

Patients with unresected breast cancer that are eligible for neoadjuvant chemotherapy that present with biopsy proven positive axillary nodes.

Study duration:

From February 2009 to February 2012 - 3 years

ELIGIBILITY:
Conditions for patient eligibility

Inclusion criteria:

* Patients must be female.
* Patients must be 18 years of age or older.
* Patients with stage IIA, IIB, IIIA (T1-3 and N1-2) breast cancer. Clinical N0 accepted if biopsy proven node disease.
* Patients that have biopsy proven positive axillary disease made by core needle biopsy or fine needle aspiration .
* Patients that accept to undergo neoadjuvant chemotherapy; patients are eligible until the day of surgery.
* Patients with bilateral breast cancer are eligible. Sentinel node biopsy is allowed on the contralateral breast if there is no disease in the axilla prior to chemotherapy.
* Patients that understand, accept and have signed the approved consent form.

Exclusion Criteria:

* Patients with inflammatory breast cancer.
* Patient with stage IIIB, IIIC or IV breast cancer (T4 and N3) Patients with clinical N3 disease are excluded.
* Patients that have had previous axillary dissection or an axillary sentinel node biopsy; (patients that have had excisional biopsy or ipsilateral tumorectomy are eligible).
* Patients that have had previous radiotherapy to the axillary nodes
* Patients that have had mammary reduction
* Patients that are medically unfit to receive chemotherapy, as evaluated by the treating physician.
* If the injection of blue dye is planned, patients with hypersensitivity or allergy to isosulfan blue, Patent blue or methylene blue or radiocolloid dye are ineligible.
* Patients who are pregnant or breast feeding .
* Psychiatric or addictive disorders or other conditions that preclude the patient from meeting the study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2009-02; Primary Completion 2012-02 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The false negative rate of sentinel node biopsy following neoadjuvant chemotherapy in biopsy proven node positive breast cancer. | 4-7 months

SECONDARY OUTCOMES:
Evaluate the accuracy of clinical evaluation and ultrasound examination in determining the presence of residual disease following neoadjuvant chemotherapy in biopsy proven node positive breast cancer. | 3-6 months
Evaluate the technical success rate of sentinel node biopsy following neoadjuvant chemotherapy | 4-7 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Boileau, MD FRCSC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre de recherche du Centre hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Boileau JF, Poirier B, Basik M, Holloway CM, Gaboury L, Sideris L, Meterissian S, Arnaout A, Brackstone M, McCready DR, Karp SE, Trop I, Lisbona A, Wright FC, Younan RJ, Provencher L, Patocskai E, Omeroglu A, Robidoux A. Sentinel node biopsy after neoadjuvant chemotherapy in biopsy-proven node-positive breast cancer: the SN FNAC study. J Clin Oncol. 2015 Jan 20;33(3):258-64. doi: 10.1200/JCO.2014.55.7827. Epub 2014 Dec 1. PMID 25452445